CLINICAL TRIAL: NCT01811719
Title: An Enhanced Nurse Home Visitation Program To Prevent Intimate Partner Violence
Brief Title: Enhanced Nurse Home Visitation to Prevent Intimate Partner Violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Portland State University (Other)
Responsible Party: Principal Investigator, Lynette Feder, Assistant Dean and Director, PAF Doctoral Program, University of Central Florida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CDC 555
Record Dates: First submitted 2013-03-08; First posted 2013-03-15 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Violence; Emotional Abuse; Pregnancy; Parenting
Keywords: Intimate Partner Physical Violence; Intimate Partner Emotional Abuse; Intimate Partner Controlling Behaivor; Pregnancy Outcomes; Quality of Parental Care Giving; Maternal Life Course
MeSH Terms: interventions — Neurofilament Proteins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced NFP (NFP+) (Experimental): Enhanced NFP(NFP+)provides for the usual NFP services plus a three-prong experimental preventive intervention:
  1. Structured and regularly occuring assessments for intimate partner violence (IPV);
  2. McFarlane and Parker Brochure Driven Intervention for women experiencing IPV, including safety planning, referrals, and advocacy; and
  3. Markman and Stanley Within My Reach Training which is a skills-based curriculum delivered to all participants focusing on improving relationship deicsions and outcomes.
  Interventions: Behavioral: Enhanced NFP (NFP+)
- NFP as usual (Active Comparator): The Nurse Family Partnership is a well-known and widely used nurse home visit program developed by David Olds. It has been rigorously tested and replicated and is now considered a best practice.
  Interventions: Behavioral: NFP as usual

INTERVENTIONS:
Behavioral: Enhanced NFP (NFP+) — Women in the experimental group received three possible interventions. First they received regular and periodic structured intimate partner violence (IPV) assessments from their nurse. Those who indicted any IPV - whether physical violence or emotional abuse or controlling behavior - were then given the Parker-McFarlane Brochure Intervention. Finally, all women were provided the Markman and Stanley Within My Reach curriculum according to their needs and interests.
  Other Names: Markman and Stanley Within My Reach Training Curriculum; McFarlane and Parker Brochure Driven Intervention
  Arms: Enhanced NFP (NFP+)
Behavioral: NFP as usual — The Nurse Family Partnership is a well-known and widely used nurse home visit program developed by David Olds. It has been rigorously tested and replicated and is now considered a best practice.
  Other Names: Nurse Family Partnership
  Arms: NFP as usual

SUMMARY:
An Enhanced Nurse Home Visitation Program To Prevent Intimate Partner Violence; This randomized trial of an intervention to assess and prevent intimate partner violence during pregnancy and the post-partum builds upon the David Olds model of nurse home visitation (Nurse Family Partnership or NFP) for high risk mothers and infants that has shown to be effective in multiple settings in preventing child abuse and enhancing maternal and child health and psychosocial outcomes. However, prior research has shown that the NFP intervention is not as effective in homes where there is intimate partner violence (IPV). Although the NFP by itself has reduced IPV in one setting, it has not in another. The proposed study will test the efficacy of an enhanced NFP intervention, the ECI or Enhanced Choice Intervention among women referred to an existing NFP program in Portland, Oregon. The ECI is based on a choice or empowerment model whereby women can choose among interventions related to her goal for her current intimate relationship. If IPV or emotional abuse or controlling behaviors are assessed, the intervention is based on two interventions shown to be effective in assessing for and reducing repeat IPV (the Sullivan Advocacy Intervention and the McFarlane and Parker brochure driven intervention). For women desiring to enhance marital quality, the Markman and Stanley PREP model that has been shown to enhance relationship quality will be offered. The PREP model also has some preliminary evidence of preventing IPV. For women with other risk factors for IPV in their own or their partners' history (e.g. exposure to parental IPV, child abuse, substance abuse), community resource linkage (beyond referral) strategies as with the NFP model will be used to obtain community resources to address these risk factors. 250 women referred to the Multnomah County Health Department will be randomized to the experimental (NFP plus ECI) or control condition (NFP) and visited according to the regular NFP schedule during pregnancy and until the infant is 24 months old. The intervention will concentrate on the prenatal and immediate (first 6 months) post partum period with regular IPV, emotional abuse and controlling behavior assessments throughout the NFP period. Baseline and outcome measurement (CTS2, WEB, TPMI, depression - Edinborough, & parenting stress), will occur at 3 months before delivery, 9 months & 21 months post-partum with multivariate MANOVA, SEM and growth curve analyses.

ELIGIBILITY:
Inclusion Criteria:

* No more than 28th week of gestation
* Low income
* Speak English or Spanish
* Pregnant with first child
* Minimum of 15 years of age at time of entrance into study

Exclusion Criteria:

* Women experiencing high risk pregnancies

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 238 (Actual)
Dates: Start 2007-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Decreased Intimate Partner Physical Violence from Baseline to Two-Year Follow-Up. | baseline, one year follow-up, and two year follow-up
  Women were given several different standardized measures regarding the amount of physical violence they might be experiencing including the Strauss Conflict Tactic Scale (CTS2r), Relationship Danger Assessment (RDA), and Proximal Antecedents of Violent Episodes Scale (PAVE).

SECONDARY OUTCOMES:
Decreased Intimate Partner Emotional Abuse & Controlling Behaviors from Baseline to Two-Year Follow-Up. | baseline, one year follow-up, and two year follow-up
  The women in the sample were given several standardized measures regarding emotional abuse and controlling behaviors including the Straus Conflict Tactic Scale (CTS2r), Psychological Maltreatment of Women Inventory (PWMI), Relationship Locus of Control (RLC), Communication Patterns Questionnaire (CPQ), and Relationship Danger Assessment (RDA).

OTHER OUTCOMES:
Improvements in the Quality of Life from Baseline to Two-Year Follow-Up. | baseline, one year follow-up, and two year follow-up
  Women were given several different standardized measures assessing their quality of life including the Quality of Life/Health and Wellbeing (SF-12), Quality of Marriage Index (QMI), Communication Patterns Questionnaire (CPQ).Edinburgh Depression Scale (EDI), Conflict Resolution Strategies (CSR), Relationship Locus of Control (RLC), Prenatal Psychosocial Profile (PPP) - Stress, Social Support, and Self-Esteem, Alcohol Use (AUDIT), Drug Use (DAST-10), Brief Child Abuse Potential Scale (CAPI), and the Parenting Stress Index (PSI).

CONTACTS AND LOCATIONS:
Overall Officials: Lynette F Feder, PhD, Principal Investigator — University of Central Florida; Phyllis Niolin, PhD, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Multnomah County Health Department, Portland, Oregon, United States

REFERENCES:
- [Derived] Li Q, Riosmena F, Valverde PA, Zhou S, Amura C, Peterson KA, Palusci VJ, Feder L. Preventing intimate partner violence among foreign-born Latinx mothers through relationship education during nurse home visiting. J Nurs Manag. 2022 Sep;30(6):1639-1647. doi: 10.1111/jonm.13565. Epub 2022 Mar 7. PMID 35174575
- [Derived] Feder L, Niolon PH, Campbell J, Whitaker DJ, Brown J, Rostad W, Bacon S. An Intimate Partner Violence Prevention Intervention in a Nurse Home Visitation Program: A Randomized Clinical Trial. J Womens Health (Larchmt). 2018 Dec;27(12):1482-1490. doi: 10.1089/jwh.2017.6599. Epub 2018 Oct 11. PMID 30311848